CLINICAL TRIAL: NCT06276699
Title: Efficacy of a Combination of Conservative Treatments Compared to Isometric Exercise on Clinical Outcomes in Patients With Cervical Radiculopathy - A Randomized Controlled Trial
Brief Title: Efficacy of a Combination of Conservative Treatments Compared to Isometric Exercise on Clinical Outcomes in Patients With Cervical Radiculopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Peradeniya (Other)
Responsible Party: Principal Investigator, T.Neeraja, Physiotherapist, Principal Investigator, University of Peradeniya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAHS
Record Dates: First submitted 2024-02-02; First posted 2024-02-26 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Conservative Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1.Isometric exercise (Placebo Comparator)
  Interventions: Procedure: 1.Isometric exercise 2.combined conservative treatment
- 2. Combined conservative treatment (Experimental)
  Interventions: Procedure: 1.Isometric exercise 2.combined conservative treatment

INTERVENTIONS:
Procedure: 1.Isometric exercise 2.combined conservative treatment — Exercise programs will be taught to patients with details by an experienced physiotherapist at the beginning of the study. Cervical Traction Patient will sit upright posture on a chair. Mechanical traction will be applied. It includes placement of a halo device around the neck, then the harness will be attached to the machine that applies traction force through-out the treatment, the device is controlled by the control panel. Intermittent mechanical traction will be applied for 10 minutes in which pull for 10 seconds and 5 seconds rest will be applied. Neural mobilization will be carried out using Butler's approach. The subject will be positioned in supine, and the median nerve will be mobilized using a slider.
  Other Names: Conservative management (Cervical traction, Neural mobilization)

SUMMARY:
This intervention study is to evaluate the efficacy of a combination of conservative treatments compared to isometric exercise on clinical outcomes in patients with cervical radiculopathy. It is a randomized, parallel, 2-arm superiority trial study. The study will be conducted at the District General Hospital in Trincomalee, where patients with cervical radiculopathy seek medical care. Patients who refer to the Department of Physical Medicine (DPM) from the Out Patients Department (OPD), orthopedic clinic and surgical clinic with a diagnosis of cervical radiculopathy or neck and arm pain (symptoms extending distal to the shoulder) will be eligible for recruitment. The study details will be explained to the subjects in the language that they best understand. Written informed consent will be obtained from the individuals who express their willingness to participate in the study, and they will sign the informed consent document accordingly.

ELIGIBILITY:
Inclusion Criteria:

* 35-60 years
* Neck pain > 3 months
* Clinical Prediction Rules - Positive Spurling's test (+) Distraction test (+) Upper limb tension test A (+) Cervical rotation on affected side < 60

Exclusion Criteria:

Presence of any signs or symptoms of medical red flags

* Less than 3(positive) items for the CPR
* Bilateral arm radiating pain
* Osteoporosis
* Tumor
* Whiplash injury
* Pregnancy woman
* Rheumatoid arthritis
* Post-surgery to cervical/thoracic spine

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Difference in pain intensity measured by Visual Analogue Scale (VAS) between combination of treatments and isometric exercises at 6-weeks post-baseline. | 2 times a week for 6 weeks
  Visual analog scale (VAS) is a measurement tool used in order to measure the pain Zero indicates no pain and 10 indicates maximum pain that patient feels

SECONDARY OUTCOMES:
Difference in cervical ROM measured by Goniometry between combination of treatments and isometric exercises at 6-weeks post-baseline. | 2 times a week for 6 weeks
  Measured by using a goniometer
Difference in functional disability measured by Neck Disability Index between combination of treatments and isometric exercises at 6-weeks post-baseline | 2 times a week for 6 weeks
  Neck disability index (NDI) will be used to measure the patient's level of disability

IPD SHARING:
Plan to Share IPD: Undecided